CLINICAL TRIAL: NCT03900351
Title: Influence of Virtual Reality Games on Knee Proprioception After Anterior Cruciate Ligament Reconstruction (ACLR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Mohammed Moustafa, Principal invsetigator, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2387594650
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Motor Activity; Proprioceptive Disorders; Balance; Distorted
MeSH Terms: conditions — Motor Activity; Somatosensory Disorders

STUDY DESIGN:
Intervention Model Description: There are two group of subjects:
  1. Group A (study group).
  2. Group B:(Control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Study group (Active Comparator): They will receive the Wii fit protocol of virtual reality games for 40 minutes, 3 times per week, for 8 weeks, in addition to the regular exercise rehabilitation protocol according to the criterion of Adams et al. (2012).
  Interventions: Procedure: Wii fit protocol of virtual reality games; Procedure: Regular exercise rehabilitation protocol
- Group B: Control group (Experimental): They will receive the regular exercise rehabilitation protocol only for 40 minutes, for 3 days per week, for 8 weeks.
  Interventions: Procedure: Regular exercise rehabilitation protocol

INTERVENTIONS:
Procedure: Wii fit protocol of virtual reality games — the Wii fit session by standing on the Wii fit board with bare feet, hands on hips and both eyes open. Pretest on Wii fit was done to make the subject familiar with the board and tasks of weight shift .
  Arms: Group A: Study group
Procedure: Regular exercise rehabilitation protocol — It will be according to the criterion of Adams et al. (2012).

SUMMARY:
Influence of virtual reality games(Wii Fit) on knee proprioception after anterior cruciate ligament reconstruction (ACLR) will be measured in 30 postoperative patients. The age of participants will be ranged from 20 to 30 years old. Subjects will be randomly assigned to Group A is the study group and Group B is the control group.

DETAILED DESCRIPTION:
Group A will receive the Wii fit protocol of virtual reality games, in addition to the regular exercise rehabilitation protocol, for 3 non-consecutive days per week, for 8 weeks , 40 minutes for each session. Group B will receive the regular exercise rehabilitation protocol only for 3 non-consecutive days per week for 8 weeks, 40 minutes for each session.

A Universal Weight and Height Scale: will be used to measure the patient's BMI.

Biodex Isokinetic Dynamometer: will be used to assess the knee proprioception of the affected operated leg at three target angles (30,45,and 60 degrees).

ELIGIBILITY:
Inclusion Criteria:

1. patients who will be in the early postoperative phase (week 2 after surgery)
2. patients with BMI less than 25, and more than 20.

Exclusion Criteria:

1. Patients with injury or operation accompanied by the ACLR as meniscectomy.
2. Patients with any deformities affecting knee joint alignment as genu valgus, genu varus, or genu recurvatum.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-07 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
knee proprioception at 30 degrees | 3 minutes
  Biodex Isokinetic Dynamometer will be used to measure knee proprioception.
knee proprioception at 45 degrees | 3 minutes
  Biodex Isokinetic Dynamometer will be used to measure knee proprioception.
knee proprioception at 60 degrees | 3 minutes
  Biodex Isokinetic Dynamometer will be used to measure knee proprioception

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan University, Jizan, Jazan Region, Saudi Arabia